CLINICAL TRIAL: NCT01226056
Title: Phase I/II Trial With Sorafenib in Combination With RAD001 Administered Orally in Patients With Advanced Solid Tumors, Selected on the Base of Molecular Targets
Brief Title: Sorafenib in Combination With RAD001 in Advanced Solid Tumors Selected on Molecular Targets
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: toxicity (protocol amendment under approval)
Sponsor: Southern Europe New Drug Organization (Other)
Collaborators: Novartis (Industry); Bayer (Industry)
Responsible Party: Scientific Director, SENDO
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S075SORD01
Record Dates: First submitted 2010-10-18; First posted 2010-10-21 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-10

CONDITIONS: Advanced Solid Tumors
Keywords: advanced solid tumors; Sorafenib (Nexavar®); RAD001 (everolimus); tumor molecular targets
MeSH Terms: interventions — Everolimus; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 in combination with sorafenib (Experimental)
  Interventions: Drug: RAD001 in combination with sorafenib

INTERVENTIONS:
Drug: RAD001 in combination with sorafenib — Phase I / Dose escalation: during the first cycle RAD001 (2.5-10 mg/day) will be administered alone, once a day, on days 1-14 to allow PK-profiling of the drug. From day 15 sorafenib administration (400-800 mg/day) twice a day will be added.
  The cycle 1 will last 6 weeks, subsequent cycles will last 4 weeks (the 2 drugs administered in combination from day 1 to day 28).
  Phase II: The drugs will be administered at the Recommended Dose and each treatment cycle will last 4 weeks.
  Other Names: RAD001 (Everolimus); Sorafenib (Nexavar®)

SUMMARY:
Sorafenib is an oral multikinase inhibitor and among its targets are several RTKs involved in tumor genesis (Raf, Flt-3, c-Kit and RET) and angiogenesis (VEGFR1, 2 and 3 and PDGFRß). Therefore sorafenib inhibits tumor growth by a dual mechanism, acting either directly on the tumor (through inhibition of Raf and Kit signaling) and/or on tumor angiogenesis (through inhibition of VEGFR and PDGFR signaling.

RAD001 is a novel derivative of rapamycin. It selectively inhibits mTOR directly blocking tumor cells by preventing tumor cell growth and proliferation and indirectly by inhibiting angiogenesis (via potent inhibition of the HIF-1 and consequently VEGF production).

Targeting mTOR in combination with sorafenib might lead to more profound effects on tumor cell biology than could be achieved through individual targeting of some proteins.

New drugs have often met only limited success since not always target pathways responsible for tumor development and growth are targeted. To overcome this problem, the specific pathways targeted by the investigators two drugs will be analyzed in each single patient before the inclusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with progressive disease of advanced solid tumours judged non suitable for standard treatment
2. Biopsiable lesion or archive tissue not older than 1 year to assess the expression of:

   * phosphorylated AKT
   * phosphorylated p70S6
   * RKIP (Raf Kinase Inhibitor Protein)
   * phosphorylated ERK1/2 The presence of at least one of the previous targets will be mandatory for patient enrolment
3. At least 1 uni-dimensional measurable lesion according to modified RECIST
4. Life expectancy of at least 12 weeks
5. Age ≥ 18 years old
6. ECOG Performance Status of 0 or 1
7. Adequate bone marrow, liver, and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to start of first dose:

   * Haemoglobin ≥9.0 g/dL (5.6 mmol/L)
   * Absolute neutrophil count (ANC)≥1.5 x 109/L
   * Platelet count ≥100 x 109/L
   * Total bilirubin ≤1.5 x upper limit of normal (ULN)
   * ALT and AST ≤2.5 x ULN (≤5 x ULN for patients with liver involvement of their cancer)
   * Alkaline phosphatase ≤4 x ULN
   * PT-INR/PTT <1.5 x ULN
   * Serum albumin levels ≥2.5 mg/dl
   * Serum creatinine ≤1.5 x ULN
8. HBV/HCV testing in the 2 weeks before treatment start in specific categories of patient with hepatitis B and C risk factors and in additional patients at the discretion of the investigators according to guidelines in Appendix 6.
9. All fertile patients must use adequate contraception while on study and for three subsequent months
10. Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to performing any study specific procedures

Exclusion Criteria:

1. History of cardiac disease: congestive heart failure (NYHA II-IV), active coronary artery disease - CAD (MI more than 6 months prior to study entry is allowed), cardiac arrhythmias requiring antiarrhythmic therapy (betablockers or digoxin are permitted) or uncontrolled hypertension
2. History of HIV infection or chronic hepatitis B or C
3. Patients with NSCLC squamous histotype
4. Recurrent hemoptysis or cerebrovascular accident within 12 months, or peripheral vascular disease with claudication on less than 1 block (about 150 metres), or history of clinically significant bleeding non-traumatic
5. Deep venous thrombosis or pulmonary embolus within 1 year or ongoing need for full-dose oral or parenteral anticoagulation
6. Clinically active infections (> Grade 2 NCI-CTC AE version 3.0)
7. Evidence of CNS tumor metastases
8. History of organ allograft
9. Pre-existing thyroid abnormality where thyroid function cannot be maintained in the normal range by medication
10. Serious, non-healing wound, ulcer, or bone fracture
11. Second malignancies within the past 5 years (except for non - melanoma skin cancer and cervical carcinoma in situ)
12. Pregnant or breast-feeding patients
13. Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
14. Any condition that is unstable or could jeopardize the safety of the patient and his/her compliance in the study
15. Patients unable to swallow oral medications
16. Any malabsorption condition
17. Prior treatment with sorafenib or m-TOR inhibitors
18. Ongoing requirement for systemic corticosteroid medication or other immunosuppressants
19. Radiotherapy within 3 weeks of start of study drug. Palliative radiotherapy is allowed. Major surgery within 4 weeks of study entry
20. Radiotherapy involving > 30% of the active bone marrow
21. Autologous bone marrow transplant or stem cell rescue within 4 months of study entry
22. Use of biologic response modifiers, such as G-CSF, within 3 week of study entry. Patients taking chronic erythropoietin are permitted provided no dose adjustment is undertaken within 2 months prior to the study or planned during the study period
23. Investigational drug therapy outside of this trial during or within 4 weeks of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose (MTD) | 6 weeks
  The maximum tolerated dose (MTD) is defined as the dose in which 2 of 3 or 2 of 6 patients experience a DLT. The Recommended Dose is identified as one dose level below the MTD.
Phase II: PFS (Progression Free survival) rate | 3 months

SECONDARY OUTCOMES:
Phase I: Pharmacokinetics profile of both drugs | 6 weeks
Phase II: overall survival | 15 months
Tumor response | every 8 weeks
  Evaluated according to RECIST criteria
Objective Response Rate (ORR) | 15 months
Incidence and severity of AEs | 36 months
  graded according to CTCAE criteria v3.0

CONTACTS AND LOCATIONS:
Overall Officials: filippo De Braud, MD, Study Chair — IEO, Milano (Italy)
Locations (1):
- Istituto Europeo di Oncologia,, Milan, Italy